CLINICAL TRIAL: NCT03416972
Title: Identification of Acute Radiation-induced Cardiac Toxicity After Non-small Cell Lung Cancer Radiotherapy With Advanced Multi-modality Imaging (RICT-LUNG)
Brief Title: Detecting Radiation-Induced Cardiac Toxicity After Non-Small Cell Lung Cancer Radiotherapy
Acronym: RICT-LUNG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: R-17-360
Record Dates: First submitted 2017-12-22; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Non-small Cell Lung Cancer; Radiation Toxicity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage I-III NSCLC patients: Stage I/II NSCLC patients receiving standard stereotactic body radiation therapy and Stage III patients receiving Standard platinum-based chemoradiotherapy will receive PET/MRI, DCE-CT, ECG/EKG, and bloodwork before and six weeks post treatment.
  Interventions: Radiation: Standard platinum-based chemoradiotherapy

INTERVENTIONS:
Radiation: Standard platinum-based chemoradiotherapy — Stage III patients: Standard platinum-based chemotherapy, total radiation dose 60 Gy in 30 fractions. Stage I/II patients: Standard radiotherapy, total radiation dose of 54 Gy in 3 fractions (peripheral), 55 Gy in 5 fractions (near chest wall), or 60 Gy in 8 fractions (central).

SUMMARY:
Lung cancer is the most common cause of cancer death in Canada. For approximately 30% of patients that present with locally-advanced non-small cell lung cancer (NSCLC), the standard treatment is curative-intent concurrent chemoradiotherapy. Outcomes remain poor, with 5-year survival of only 20%. Despite the long-held belief that higher radiation doses lead to improved overall survival (OS), the landmark randomized trial (RTOG 0617) showed the opposite. The investigators hypothesize that the inferior survival observed may be due to unexpected heart toxicity as secondary analysis revealed that the heart dose was a strong predictor of inferior OS. Up to now, change in heart function is typically detected histologically, requiring autopsy tissue. Therefore, a non-invasive marker of early heart damage is required. Hybrid PET-MRI has become available in Canada only recently. The ability to simultaneously perform metabolic imaging with functional and tissue imaging allows for novel assessment of heart toxicity. The primary objective is to examine the utility of hybrid PET-MRI and DCE-CT to assess acute changes in heart function and to measure inflammation before, and six weeks after NSCLC radiotherapy. A pilot of 20 patients with Stage I-III NSCLC will be enrolled. The findings of this study will aid in the design of new studies to reassess dose escalation for locally advanced NSCLC while limiting the risk of heart toxicity. FDG PET will be used to simultaneously assess both cardiac inflammation and tumour response. Quantitative DCE-CT will also be used to measure ventilation and perfusion changes in the normal lung and tumour after radiotherapy, providing image data that can comprehensively assess both tumour response and potential toxicity in both the heart and lungs. Such information is crucial in understanding the disease and its response to treatment. This data will also aid in the design of radiation techniques that spare the heart in other patients with any thoracic malignancies, including breast cancer, lymphoma, and esophageal cancer.

DETAILED DESCRIPTION:
The investigators propose a longitudinal imaging pilot study composed of 20 Stage I-III NSCLC patients before, and six weeks after standard radiotherapy using a hybrid 3T-PET/MRI system (Biograph mMR, Siemens Healthcare) and a GE Revolution 256-slice CT scanner. The imaging protocol is designed to detect acute changes in myocardial perfusion, inflammation, edema, left ventricular ejection fraction, normal lung and tumour perfusion, and tumour metabolism. During each imaging session, patients will receive an 18F-FDG PET scan to image macrophage-related inflammation and tumour metabolism, MRI to identify edema, mature fibrosis or scar, and Dynamic contrast enhanced CT (DCE-CT) imaging to image perfusion and (LVEF). All images will be fused and rendered with radiation treatment planning dose distributions. Parameters such as Standard Uptake Value (SUV) will be used to compare PET scans, while heart volume and presence of Gadolinium enhancement will be used to compare MRI scans. Blood flow, blood volume, and permeability will be used to compare CT scans. Blood tests including Erythrocyte Sedimentation Rate (ESR), high sensitivity C-reactive protein, and troponin at each timepoint will also be performed to detect cardiac inflammation. Comparisons between Stage I/II and Stage III patients will allow us to determine whether our metrics for heart changes is radiation related. Relative differences from the six-week time point to baseline will be correlated with the radiation dose distribution to attempt to define a dose-response relationship between radiation dose and cardiac toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Ability to provide informed consent
* Histologically confirmed carcinoma of the lung
* Stage I-III NSCLC
* Stage I-II patients to receive 54 Gy in 3 fractions, 55 Gy in 5 fractions, or 60 Gy in 8 fractions (treated every other day)
* Stage III patient to receive concurrent chemoradiation ( 60 Gy in 30 daily fractions)
* No prior RT to the thorax
* ECOG performance status 0-1 within one month of accrual
* Expected lifespan at least 1 year
* Negative pregnancy test within one month of accrual if woman is premenopausal
* Patient presented at multidisciplinary tumor board or quality-assurance rounds
* Satisfactory pulmonary function tests as determined by the treating radiation oncologist (ie. FEV1 >= 0.8 for Stage III NSCLC and no threshold for Stage I/II).

Exclusion Criteria:

* Patients receiving Prescription RT dose to anything other than LRCP standards for Stage I-III NSCLC.
* Prior history of atrial fibrillation
* Previous coronary bypass surgery
* Patients with severe reversible airways obstruction
* Patients with acute coronary syndrome (STEMI/non-STEMI and unstable angina)
* AV block without pacemaker
* Patients who are renal insufficient (eGFR <40)
* Patients with asthma
* Allergy to iodinated contrast for scans (study subject will be eligible for non-contrast scans)
* Use of metformin-containing products less than 24 hours prior to CT contrast administration
* Other contraindications to iodinated contrast media as determined by the research team.
* Allergy to gadolinium for scans using contrast; will be eligible for non-contrast scans.
* Other contraindications to gadolinium contrast media as determined by the research team.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ultimately, the sample size was based upon practical considerations and that 20 NSCLC patients (10 Stage I/II and 10 Stage III) could be accrued relatively easily from new patient clinics, while sufficiently providing enough evidence to validate the imaging techniques to be used as a non-invasive measure for future clinical trials aimed at reducing or mitigating radiation-induced cardiac toxicity.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Detection of Imaging Biomarkers of acute cardiac inflammation | 6 weeks
  FDG-PET imaging to detect increase in cardiac inflammation compared to baseline with corresponding blood markers (Erythrocyte Sedimentation Rate (ESR), high sensitivity C-reactive protein, and troponin levels in blood (inflammation)).
Detection of Imaging Biomarkers of acute cardiac perfusion changes | 6 weeks
  DCE-CT imaging to detect changes in acute cardiac perfusion changes compared to baseline.
Detection of Imaging Biomarkers of acute changes in Left-ventricular ejection fraction (LVEF) | 6 weeks
  Contrast-enhanced CT imaging to detect acute changes in LVEF compared to baseline.
Detection of cardiac fibrosis | 6 weeks
  Gadolinium Enhanced MR imaging to detect cardiac fibrosis compared to baseline

SECONDARY OUTCOMES:
Tumour Response (metabolism) | 6 weeks
  FDG-PET imaging to detect tumour metabolism changes compared to baseline.
Tumour Response (perfusion) | 6 weeks
  DCE-CT imaging to detect changes in tumour perfusion compared to baseline
Acute Changes in Lung Ventilation | 6 weeks
  4D-CT imaging to detect changes in lung ventilation compared to baseline
Acute Changes in Lung Perfusion | 6 weeks
  DCE-CT imaging to detect changes in lung perfusion compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Gaede, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No